CLINICAL TRIAL: NCT00266344
Title: MK0928 Phase IIb Dose-range Finding Study -Primary Insomnia
Brief Title: MK0928 Study in Adult Patients With Primary Insomnia (0928-040)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Executive Vice President, Clinical and Quantitative Sciences, Merck & Co., Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0928-040; MK0928-040; 2005_106
Record Dates: First submitted 2005-12-14; First posted 2005-12-16 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Primary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — gaboxadol; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0928, gaboxadol / Duration of Treatment 3 Weeks
Drug: Placebo / Duration of Treatment 3 Weeks

SUMMARY:
A study to evaluate the efficacy, safety and tolerability of MK-0928 in Primary Insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of primary insomnia

Exclusion Criteria:

* Patients with an active psychiatric disorder other than primary insomnia

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 520
Dates: Start 2005-11; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Patient-reported total sleep time.

SECONDARY OUTCOMES:
Patient-reported time to sleep onset, number of awakenings, wake time after sleep onset and premature awakening.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC